CLINICAL TRIAL: NCT04135690
Title: Hepatic Arterial Infusion Chemotherapy Plus Toripalimab Versus Hepatic Arterial Infusion Chemotherapy Plus Sorafenib for Hepatocellular Carcinoma With Portal Vein Tumor Thrombus: a Non-comparative, Prospective, Randomized Trial
Brief Title: HAIC Plus Toripalimab vs. HAIC Plus Sorafenib for HCC With PVTT: a Non-comparative, Prospective, Randomized Trial
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Shi Ming, Proffessor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S0905
Record Dates: First submitted 2019-10-20; First posted 2019-10-23 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Hepatic arterial infusion chemotherapy; Oxaliplatin, 5-Fluorouracil and Leucovorin; Toripalimab; Sorafenib
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — toripalimab; Sorafenib; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HAIC plus toripalimab (Experimental): Hepatic arterial infusion of oxaliplatin , fluorouracil, and leucovorin every 3 weeks. Toripalimab 240mg intravenously every 3 weeks.
  Interventions: Procedure: Hepatic arterial infusion chemotherapy; Drug: Toripalimab
- HAIC plus sorafenib (Active Comparator): Hepatic arterial infusion of oxaliplatin , fluorouracil, and leucovorin every 3 weeks. Sorafenib 400mg twice daily (Bid) oral dosing.
  Interventions: Procedure: Hepatic arterial infusion chemotherapy; Drug: Sorafenib
- Patients receiving TKI plus ICI (Other): Patients, who meet the inclusion criteria but withdraw consent or reject this study, receive systemic treatment according to the doctor. Systemic treatment include atezolizumab+bevacizumab, camrelizumab+apatinib, sintilimab+bevacizumab and so on.
  Interventions: Drug: systemic treatment

INTERVENTIONS:
Procedure: Hepatic arterial infusion chemotherapy — administration of oxaliplatin , fluorouracil, and leucovorin via the tumor feeding arteries every 3 weeks
  Arms: HAIC plus sorafenib; HAIC plus toripalimab
Drug: Toripalimab — 240mg intravenously every 3 weeks
  Arms: HAIC plus toripalimab
Drug: Sorafenib — 400mg bid po
  Arms: HAIC plus sorafenib
Drug: systemic treatment — atezolizumab+bevacizumab, camrelizumab+apatinib, sintilimab+bevacizumab and so on
  Arms: Patients receiving TKI plus ICI

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of hepatic arterial infusion chemotherapy of oxaliplatin, 5-fluorouracil and leucovorin plus toripalimab versus hepatic arterial infusion chemotherapy of oxaliplatin, 5-fluorouracil and leucovorin plus sorafenib in patients with hepatocellular carcinoma (HCC) with portal vein tumor thrombus.

DETAILED DESCRIPTION:
Our previous study showed that hepatic arterial infusion chemotherapy (HAIC) of oxaliplatin, 5-fluorouracil and leucovorin plus sorafenib was more effective and safe than sorafenib for hepatocellular carcinoma with portal vein tumor thrombus. Programmed cell death protein-1 (PD-1) antibody was effective and tolerable in patients with advanced hepatocellular carcinoma. No study has compared HAIC plus toripalimab with HAIC plus sorafenib. Thus, the investigators carried out this prospective, randomized, non-comparative study to find out it.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of HCC was based on the diagnostic criteria for HCC used by the European Association for the Study of the Liver (EASL)
* Patients must have at least one tumor lesion that can be accurately measured according to EASL criteria.
* Patients with portal vein tumor thrombus
* Eastern Cooperative Oncology Group performance status of 0 to 2
* With no previous treatment
* No Cirrhosis or cirrhotic status of Child-Pugh class A only
* Not amendable to surgical resection ,local ablative therapy and any other cured treatment.
* The following laboratory parameters:

Platelet ≥75,000/μL Hemoglobin ≥ 8.5 g/dL Total bilirubin ≤ 30mmol/L Serum albumin ≥ 32 g/L ASL and AST ≤ 5 x upper limit of normal Serum creatinine ≤ 1.5 x upper limit of normal INR ≤ 1.5 or PT/APTT within normal limits Absolute neutrophil count (ANC) >1,500/mm3

• Ability to understand the protocol and to agree to and sign a written informed consent document

Exclusion Criteria:

* Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy
* Known history of HIV
* History of organ allograft
* Known or suspected allergy to the investigational agents or any agent given in association with this trial.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Evidence of bleeding diathesis.
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.
* Known central nervous system tumors including metastatic brain disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-10-20 (Actual); Primary Completion 2023-12-20 (Estimated); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
Progression free survival rate at 6 months | 6 months
  Progression was defined as progressive disease by independent radiologic review according to RECIST or death from any cause

SECONDARY OUTCOMES:
Overall survival (OS) | 6 months
  OS is the length of time from the date of randomization until death from any cause.
Progression free survival (PFS) | 6 months
  PFS is defined as the time from the date of randomization to the date of the first objectively documented tumor progression or death due to any cause.
Objective response rate (ORR) | 6 months
  ORR, as determined based on tumor response according to RECIST 1.1, is defined as the proportion of all randomized subjects whose best overall response (BOR) is either a CR or PR.
Adverse events | 6 months
  Safety will be evaluated according to the NCI CTCAE Version 4.03. All observations pertinent to the safety of the study medication will be recorded on the CRF and included in the final report.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Center Sun Yat-sen University, Guangzhou, Guangdong, China